CLINICAL TRIAL: NCT03030989
Title: A Double-blind Randomized Placebo Controlled Clinical Trial Evaluating Effect of Chlorhexidine Gluconate 2% Cloth vs Placebo Cloth Baths on the Incidence of Central Line-Associated Blood Stream Infections in Outpatient Hematopoietic Stem Cell Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB16-1059
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Stem Cell Transplant Complications
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine Gluconate 2% Wipe (Active Comparator)
  Interventions: Drug: Chlorhexidine Gluconate 2% Wipe
- Placebo wipe (Placebo Comparator)
  Interventions: Drug: Placebo Wipe

INTERVENTIONS:
Drug: Chlorhexidine Gluconate 2% Wipe
  Arms: Chlorhexidine Gluconate 2% Wipe
Drug: Placebo Wipe
  Arms: Placebo wipe

SUMMARY:
This study evaluates the use of 2% CHG washcloths in an outpatient setting for adults after hematopoietic stem cell transplant in prevention of central line associated blood stream infections. Half of the participants will use 2% CHG washcloths and other half will use placebo washcloths.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the University of Chicago Hematopoietic Stem Cell Transplant Unit for transplant
* Age 18 and up

Exclusion Criteria:

* Experienced an allergy or rash related to use of chlorhexidine washcloths or other chlorhexidine products
* Extensive open wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01-02 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorhexidine Gluconate 2% Wipe: Chlorhexidine Gluconate 2% Wipe
- Placebo Wipe: Placebo Wipe
Period: Overall Study
Arm/Group | Chlorhexidine Gluconate 2% Wipe | Placebo Wipe
Started | 21 | 29
Completed (Dropout due to fatigue at using wipes was high; compliance is enhanced with monitoring in hospital.) | 9 | 15
Not Completed | 12 | 14
Not completed — Fever | 2 | 2
Not completed — Rash | 2 | 1
Not completed — Fatigue/Overwhelmed | 1 | 5
Not completed — Positive Blood Cultures | 2 | 1
Not completed — Line Removed | 0 | 2
Not completed — No longer interested | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Gluconate 2% Wipe | Placebo Wipe | Total
Number analyzed (Participants) | 21 | 29 | 50
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 75] | 61 [23 to 74] | 61.5 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 11 | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 28 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 14 | 23 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 29 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Blood Stream Infections
Description: Blood stream infections are defined by the presence of bacteria in the blood
Time Frame: 14 weeks
Population: Among all subjects enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate 2% Wipe | Placebo Wipe
Number analyzed (Participants) | 21 | 29
Participants | 1 | 2

2. Primary Outcome: Number of Participants With Clinical (Culture-negative) Sepsis
Description: Clinical (culture-negative) sepsis is defined by the presence of low blood pressure without bacteria in the blood
Time Frame: 14 weeks
Population: Among all subjects enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate 2% Wipe | Placebo Wipe
Number analyzed (Participants) | 21 | 29
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Chlorhexidine Gluconate 2% Wipe | Placebo Wipe
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/29
Other Adverse Events (participants affected / at risk) | 2/21 | 1/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorhexidine Gluconate 2% Wipe (N=21) | Placebo Wipe (N=29)
Rash (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT03030989/Prot_SAP_000.pdf